CLINICAL TRIAL: NCT01836978
Title: Prehabilitation to Enhance Postoperative Functional Capacity Following Radical Cystectomy: Combining Physical Exercise to Stress Reduction Strategies and Nutritional Supplementation
Brief Title: Prehabilitation to Enhance Postoperative Functional Capacity Following Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Franco Carli, MD, MPhil, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-454-SDR
Record Dates: First submitted 2013-04-09; First posted 2013-04-22 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Bladder Cancer; Entire Ileal Conduit; Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients in this group will follow standard MUHC clinical guidelines. This group will receive general instructions, by the preoperative clinic nurse, on exercises (breathing, ankle rotation) to be done before and after surgery. They will also be seen by a nutritionist who will provide general counseling for healthy eating.
- Prehabilitation (Experimental): Patients in this group will follow the multimodal protocol consisting of nutritional counseling with Immunocal® whey protein supplementation, an individualized physical exercise program, and stress reduction strategies.
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — Patients in this group will follow the multimodal protocol consisting of nutritional counseling with Immunocal® whey protein supplementation, an individualized physical exercise program and stress reduction strategies.
  Arms: Prehabilitation

SUMMARY:
The process of enhancing the functional capacity of an individual before an operation to enable him or her to withstand the stress of surgery has been termed prehabilitation. It has been shown that poor baseline capacity for physical performance and poor nutritional status increase the risk of complications after major non cardiac surgery and prolong recovery. A controlled randomized study in patients undergoing radical cystectomy for cancer is therefore proposed to determine the impact of multimodal prehabilitation on functional exercise capacity and functional recovery. Patients who accept to be enrolled in the study will be randomized to either a group receiving a multimodal intervention which includes nutritional supplementation (Immunocal® whey protein) combined with a physical exercise program and stress reduction strategies before and after surgery, or a control group who will receive standard preoperative treatment as per our institution.

DETAILED DESCRIPTION:
Study Arms

1. Standard group Patients in this group will follow standard MUHC clinical guidelines. This group will receive general instructions on exercises (breathing, ankle rotation) to be done before and after surgery by the preoperative clinic nurse. They will also be seen by a nutritionist who will provide general counseling for healthy eating.
2. Prehabilitation group Patients in this group will follow the multimodal protocol consisting of nutritional supplementation, a specific physical exercise program and stress reduction strategies.

Randomization Patients will be assigned to the two groups using a computer-generated randomization process whereby brown sealed envelopes will be prepared and opened after patients' consent has been signed.

Components of prehabilitation

1. Nutritional supplementation The nutritional status of patients affected by bladder cancer is directly influenced by the presence of cancer which has an impact on all aspects of intermediary (protein, carbohydrate, lipid, trace element, vitamin) metabolism, and by other factors such as age, adjuvant cancer therapy and stage of the disease. In addition, a patient who is undernourished before surgery has greater risk of morbidity and mortality. The primary goal of nutrition therapy during the perioperative period is thus to optimize nutrient stores pre-operatively and provide adequate nutrition to compensate for the catabolic response of surgery postoperatively. This includes preventing the loss of lean body mass which is inversely correlated with the survival of critically ill patients.

   The patients' nutritional status and adequacy of dietary intake will be assessed by a nutritionist using a three day food record and the Subjective Global Assessment tool. Percentage of lean body mass and fat will be measured with bioelectrical impedance. Serum albumin will also be measured. All patients in the prehabilitation group will be provided with a whey protein supplement (Immunocal®, Immunotec Inc.) and will be provided with strategies to optimize dietary energy and protein intake. The quantity of supplement the patient will be required to consume daily will depend on the estimated deficit in dietary protein intake. This will be determined based on the difference between usual protein intake and protein requirement, as assessed by the nutritionist at the baseline assessment. Patients in the control group will receive general instructions about healthy eating.

   Compliance will be monitored weekly through phone calls by the study coordinator. The patients will also be asked to complete a journal detailing the quantity of nutritional supplement consumed each day.
2. Physical exercise program It has been shown that prehabilitation can improve postoperative physical function in cancer patients undergoing colorectal surgery and lung resection, and these changes are associated with improvements in mental health, vitality, and self-perceived health. Moreover, it appears that subjects whose fitness deteriorated preoperatively have more surgical complications and require intensive care. A recently published systematic review of preoperative physical exercise by Valkenet et al reported less postoperative complications and shorter length of stay in abdominal surgery patients. Although the role of exercise intensity is unclear, it appears that moderate exercise, carried out in a combination of aerobic and resistance training components, is sufficient to build adequate physiological reserve and energy, even in patients who receive chemotherapy.

The exercise component will consist of approximately 60 min of resistance and aerobic training, for a minimum of 3 days per week. The exercise program will be individualized based upon the baseline fitness test (according to the American College of Sport Medicine, ACMS, standard) and will include: a 5 min warm-up, either 25 min of aerobic exercise (starting at 30- 40 % of heart rate reserve, HRR), and 25 min of resistance training (8 exercises targeting major muscle groups performed at moderate intensity), and a 5-10 min cool-down and stretching period. All exercises will be clearly explained and demonstrated by the kinesiologist at baseline. Patients will be asked to carry out this program at home, unsupervised, but will be monitored with weekly telephone calls. Training intensity progression will occur when the participant can complete aerobic exercise on mild exertion and/or when the participant can complete 15 repetitions of a given resistance exercise. Participants will be provided with resistance bands and an exercise mat, as well as a pedometer and a heart rate monitor, which can be used by the participant to monitor progress and by the kinesiologist to monitor daily compliance. A log book will also be completed to report all activities and frequency of exercises completed.

The kinesiologist will follow all the participants on a weekly basis to ensure program compliance and address any barriers that may prevent ongoing participation.

The control group will receive general instructions on how to exercise during hospital stay while in bed, walking and sitting.

C. Anxiety reduction strategy.

It is expected that patients undergoing bladder surgery for cancer are anxious and depressed. The control group will receive general instructions in the preoperative clinic about the perioperative care and breathing exercises, while those in the prehabilitation group will be seen by a psychologist coordinator who will provide different strategies to deal with anxiety and depression (guided imagery, relaxation, visualization, yoga).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and older
* Referred electively for radical resection of a bladder tumor (may or may not receive adjuvant therapy).

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) health status class 4-5 or co-morbid medical, physical and mental conditions (e.g. dementia, disabling orthopedic and neuromuscular disease, psychosis)
* Severe cardiac abnormalities
* Severe end-stage organ disease such as cardiac failure (New York Heart Association classes I-IV)
* Chronic Obstructive Pulmonary Disease (COPD)
* Hepatic failure (liver enzymes >50% over the normal range)
* Sepsis
* Morbid obesity (BMI >35)
* Anemia (hematocrit < 30 %, haemoglobin <100 g/L, albumin < 25 g/L)
* Poor comprehension of English or French.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Six minute walking test (6MWT) | up to 8 weeks after surgery
  The 6MWT evaluates the ability of an individual to maintain a moderate level of physical activity over a time period reflective of the activities of daily living. Subjects are instructed to walk back and forth, in a 20 m stretch of hallway, for six minutes, at a pace that would make them tired by the end of the walk

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, MD, Principal Investigator — Perioperative Programme (POP)
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Li C, Carli F, Lee L, Charlebois P, Stein B, Liberman AS, Kaneva P, Augustin B, Wongyingsinn M, Gamsa A, Kim DJ, Vassiliou MC, Feldman LS. Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study. Surg Endosc. 2013 Apr;27(4):1072-82. doi: 10.1007/s00464-012-2560-5. Epub 2012 Oct 9. PMID 23052535